CLINICAL TRIAL: NCT07299474
Title: Efficacy Of Lavender Aromatherapy on Anxiety and Pain Reduction During Awake Otolaryngologic Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ankona Ghosh, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004415
Record Dates: First submitted 2025-11-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Inferior Turbinate Hypertrophy; Chronic Rhinosinusitis (CRS); Rhinitis, Vasomotor; Thyroid Nodules; Vocal Fold Immobility
Keywords: Aromatherapy; Otolaryngology; Awake procedure
MeSH Terms: conditions — Rhinitis, Vasomotor; Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Aromatherapy (Experimental): Participants will be exposed to lavender aromatherapy on a cotton ball prior to procedure, and then with a diffuser during the duration of the procedure
  Interventions: Other: Lavender Aromatherapy
- Placebo (Placebo Comparator): Participants will be exposed to placebo odorless liquid, on a cotton ball prior to procedure, and then with a diffuser during the duration of the procedure
  Interventions: Other: Placebo Aromatherapy

INTERVENTIONS:
Other: Lavender Aromatherapy — Lavender essential oil on cotton ball, and in aromatherapy diffuser
  Arms: Lavender Aromatherapy
Other: Placebo Aromatherapy — Saline on cotton ball and in aromatherapy diffuser
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of lavender aromatherapy in adult patients undergoing awake otolaryngologic procedures in the outpatient clinic setting. The main questions it aims to answer are:

* Does lavender aromatherapy help reduce anxiety and/or pain, and improve patient comfort during awake otolaryngologic procedures in the clinic?
* Do patients subjectively find aromatherapy relaxing and/or beneficial during the procedure?

Researchers will compare lavender aromatherapy to placebo (an odorless liquid) to see if lavender aromatherapy helps improve patient comfort during their awake procedure

Participants will:

* Have their scheduled procedure performed with lavender aromatherapy or placebo during the duration of the procedure
* Take a short, less than 1 minute questionnaire both before and after the procedure, describing their levels of anxiety, pain and subjective impressions of the aromatherapy

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old undergoing awake otolaryngologic procedures in the outpatient clinic
* Able to provide informed consent

Exclusion Criteria:

* Hypersensitivity to fragrances
* Taking systemic NSAIDs or other systemic pain-relieving medications within 48 hours
* Taking anxiolytics, hypnotics, sedating antihistamines, antidepressants on regular basis within 4 weeks
* Pregnant or breastfeeding
* Participation in another clinical research study within the prior 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in visual analog scale anxiety, measured on a 10 cm scale | Baseline, Periprocedural and Immediately after the procedure
  A 10 cm visual analog scale is widely utilized to measure procedural anxiety, rated from 0 to 10, with 10 being the highest level of anxiety. The patient will provide a vertical mark above their level of anxiety. This number measured in mm (0-100) will be recorded both immediately before the procedure, and after the procedure, where the patient will record their average level of anxiety during the procedure. The change between pre-procedure, and post-procedure, will be recorded for each patient and compared between the lavender aromatherapy and placebo groups. The mean and median pre-procedure and post-procedure values will also be compared between the groups.
Likert scale of pain, measured on a scale of 0-10 | Immediately after the procedure
  Patients will be asked to rate their your average level of pain on a scale of 0 (no pain) to 10 (worst possible pain) on a post-procedural questionnaire
Likert scale subjective improvement with pain, measured on scale of 1-5 | Immediately after the procedure
  Patients will be asked in post-procedural questionnaire if they felt the aromatherapy helped with pain during the procedure, on a scale of 1 (strongly disagree) to 5 (strongly agree)

SECONDARY OUTCOMES:
Subjective Impressions of Lavender Aromatherapy, measured on Likert scale and in Yes/No format in post-procedural questionnaire | Immediately after the procedure
  Patients will be asked in a post-procedural questionnaire their subjective impressions of the lavender aromatherapy or placebo. The questions will be outlined as below:
  Did you feel the aromatherapy was calming during the procedure?
  1 2 3 4 5 (1 = strongly disagree, 5 = strongly agree)
  Did you find the scent pleasant? 1 2 3 4 5 (1 = strongly disagree, 5 = strongly agree)
  Do you use aromatherapy or essential oils regularly? Yes No
  Have you ever used aromatherapy or essential oils in the past? Yes No
  How likely are you to recommend the aromatherapy for future patients undergoing awake procedures?
  1 2 3 4 5 (1 = strongly disagree, 5 = strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Ankona Ghosh, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center Otolaryngology Clinics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers in order to protect patient privacy, as these patients will be undergoing awake procedures at only 1 location, and thus their results may be identified even after anonymization or de-identification.

REFERENCES:
- [Background] Braden R, Reichow S, Halm MA. The use of the essential oil lavandin to reduce preoperative anxiety in surgical patients. J Perianesth Nurs. 2009 Dec;24(6):348-55. doi: 10.1016/j.jopan.2009.10.002. PMID 19962101
- [Background] Kothari DS, Nieri CA, Tanenbaum ZG, Linker LA, Rangarajan SV. Mind-Body Therapies in the Management of Otolaryngologic Disease: A State-of-the-Art Review of Randomized Controlled Trials. Otolaryngol Head Neck Surg. 2024 Jan;170(1):45-60. doi: 10.1002/ohn.523. Epub 2023 Sep 15. PMID 37712305
- [Background] Grunebaum LD, Murdock J, Castanedo-Tardan MP, Baumann LS. Effects of lavender olfactory input on cosmetic procedures. J Cosmet Dermatol. 2011 Jun;10(2):89-93. doi: 10.1111/j.1473-2165.2011.00554.x. PMID 21649812
- [Background] Wotman M, Levinger J, Leung L, Kallush A, Mauer E, Kacker A. The Efficacy of Lavender Aromatherapy in Reducing Preoperative Anxiety in Ambulatory Surgery Patients Undergoing Procedures in General Otolaryngology. Laryngoscope Investig Otolaryngol. 2017 Nov 8;2(6):437-441. doi: 10.1002/lio2.121. eCollection 2017 Dec. PMID 29299520